CLINICAL TRIAL: NCT01975129
Title: A Pharmacokinetic Study of Vaginally and Intravenously Administered Oxytocin in Postmenopausal Women With Vaginal Atrophy
Brief Title: A Pharmacokinetic Study of Vaginally and Intravenously Administered Oxytocin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PepTonic Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXYPEP003
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Vaginal Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vagitocin (Oxytocin) (Experimental)
  Interventions: Drug: Vagitocin

INTERVENTIONS:
Drug: Vagitocin
  Other Names: Oxytocin gel 400 International Units

SUMMARY:
This study aims to evaluate the uptake of oxytocin following intravaginal administration of Vagitocin 400IU over a period of 15 days and also to compare oxytocin bioavailability after vaginal and intravenous administration. 12 healthy postmenopausal female volunteers, 40 to 70 years old with vaginal atrophy will be included and will self-administer Vagitocin intravaginally on day 2-14 (day 1 and 15 Vagitocin is given in the clinic). On day 22 a single intravenous dose of oxytocin 10 IU Syntocinon® will be given. Oxytocin plasma levels after intravaginal and intravenous administration will be analysed day 1, 15 and 22 at timepoints: -1.0, -0.5, 0, 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 5.0, 6.0 and 8.0 hours, relative to dosing. Based on the obtained plasma levels for oxytocin, pharmakokinetic variables will be calculated. The % of oxytocin which was absorbed following vaginal administration (bioavailability)will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women with vaginal atrophy as judged by the investigator
* Willing to participate in the study as indicated by signing the informed consent
* Healthy post-menopausal women between the ages of 40 and 70 years, inclusive
* Body mass index (BMI) less than or equal to 32 kg/m2 but greater than or equal to 19 kg/m2
* Judged by the Investigator to be healthy on the basis of medical evaluation

Exclusion Criteria:

* Hospitalized subjects
* Symptoms of any significant acute illnesses at the screening visit
* History of significant allergies (including food, asthma, or drug allergies including allergies to any ingredient of the trial product)
* Known history of sensitivity to oxytocin or related derivatives
* Follicle-stimulating hormone level < 40 pmol/mL
* Known history of narcotic addiction, drug abuse or alcoholism
* Simultaneously participate in another clinical study
* Use of any sex steroids including phytoestrogens, hormonal intrauterine device or herbal medicinal products with known estrogenic effects within 3 months prior to baseline
* Uncontrolled hypertension and/or hypercholesterolemia

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Oxytocin plasma levels | Day 1 to 26
  Oxytocin plasma levels after intravaginal and intravenous administration

CONTACTS AND LOCATIONS:
Overall Officials: Aino Fianu Jonasson, MD Ass Prof, Principal Investigator — Karolinska University Hopsital, Womens Health
Locations (1):
- Women's health clinic, Stockholm, Huddinge, Sweden